CLINICAL TRIAL: NCT05959122
Title: IRON DEFICIENCY ANEMIA IN RELATION TO PINCH STRENGTH AND HAND DEXTERITY IN PRESCHOOL CHILDREN
Acronym: IDA
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Essam ELDIN ABDALLAH AMER, Physical therapist at Zagazig General Hospital, El Sharkia, Egypt., Cairo University
Other Study IDs: No: P.T.REC/012/001850
Record Dates: First submitted 2023-07-15; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia, pinch strength, dexterity, preschooler children
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- group A: group (A) thirty-six non-anemic children
  Interventions: Diagnostic Test: CBC serum iron serum ferritin
- group B: group (B) twenty five children with mild IDA
  Interventions: Diagnostic Test: CBC serum iron serum ferritin
- Group C: group (C) 26 children with moderate
  Interventions: Diagnostic Test: CBC serum iron serum ferritin

INTERVENTIONS:
Diagnostic Test: CBC serum iron serum ferritin — 1. Fully automated blood cell counter (sysmex-Xs 800i) and AU 480-Chemistry auto-analyzer (Beckman Coulter Diagnostics-USA) was used for measurement of hemoglobin and serum iron levels
  2. Chemiluminescence assay using an Abbott i2000SR analyser was used to measured serum ferritin
  Other Names: measure tip to tip and tripod pinch strength by Baseline mechanical Pinch gauge (0-60 lb.) and BOT-2 used to assess manual dexterity

SUMMARY:
Anemia is a major public health problem among preschool-aged children. The evidence demonstrated that early childhood anemia is a strong predictor of adulthood anemia (Gessner, 2009). According to Egypt's Demographic and Health Survey (EDHS), prevalence rates of anemia in children aged 6-59 months ranged from 23% to 45% (EDHS, 2014). It is assumed that 50% of the cases of anemia are due to ID (Aref and Khalifa, 2019). The major health problem in Egypt is ID that affects 41.2% of children aged <5years (El-Asheer et al., 2021). The total prevalence of IDA in the Nile Delta region was 17.19% of the children (El-Shanshory et al., 2021). Iron is a trace element that is essential to form hemoglobin in red blood cells and to carry oxygen to peripheral tissues. In addition, iron plays essential functions in the mitochondria, which are crucial for regulating energy metabolism in the skeletal muscle (Kang and Li, 2012). And low iron levels limit oxygen bioavailability in the peripheral tissues, including skeletal muscle (Jolly et al., 2001).Yu-mi et al., (2020) found a low handgrip strength in anemic patients. Also, ID can impaired brain energy metabolism, along with hypo-myelination and impaired dopamine signaling, is consistently described as one of the mechanistic causes of the neurodevelopmental deficits associated with early-life ID (Thomas et al., 2020).

HYPOTHESES:

There is a relation between IDA and pinch strength and hand dexterity in preschool children.

RESEARCH QUESTION:

Is there a relation between IDA and pinch strength and hand dexterity in preschool children?

The purpose of the current study is to find the relation between IDA and:

1. Pinch grip strength (tripod and tip to tip grip strength).
2. Hand dexterity in preschool children.

DETAILED DESCRIPTION:
i. Instrumentations for selection:

1. Fully automated blood cell counter. A complete blood count (CBC) is one of the most commonly and routinely done laboratory tests It will be obtained through the use of fully automated blood cell counter (sysmex-Xs 800i).
2. Beckman coulter-AU 480- blood chemistry auto-analyzer. It is the ideal primary chemistry analyzer for measurement of the amount of serum iron in the blood. ii. Instrumentations for assessment:

Updated 23/11/12

4

1. Baseline mechanical Pinch gauge (0-60 lb.) used to measure tripod pinch strength of dominance and non-dominance hands for all participated children.
2. Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) The Bruininks-Oseretsky Test of Motor Proficiency is a standardized, norm-referenced measure

Inclusion Criteria:

1. Their age will be ranged from 5-6 years
2. The fifty anemic children will have microcytic hypochromic anemia: their Hb < 11.5 g/L (Hb from 11.0-11.4 is mild anemia and in moderate anemia Hb is from 8.0-10.9 (WHO, 2011). The serum iron is below 60 mcg/dL (Elngar et al., 2021). The Ferritin level

   <12 µg/L for children in absence of infection (WHO, 2017). ( Appendix I).
3. They will be right handed.
4. They had no history of previous hand injuries, surgeries or other functional hand limitation.
5. All children will able to follow instructions and understand commands given during test procedures.
6. Their body mass index (BMI) will be ranged from 15.2 to 15.5 kg/m2 (WHO, 2007). (Appendix II).

B. Exclusion Criteria:

Children will exclude if they have:

1. Congenital or acquired deformity in the joints of upper limb.
2. Unhealed fracture in upper limb bones.
3. Systematic disease that cause anemia such as renal or hepatic failure or a history of bone disease.
4. Blood transfusion within 3 months before measuring the hematological indices.
5. Documented trauma in the previous 12 months in the muscle fibers, or those taking medication that affecting strength.
6. Children begin with musculoskeletal problems or neurological disorders that affected their upper extremities

ELIGIBILITY:
Inclusion Criteria

1. Their age will be ranged from 5-6 years
2. The fifty anemic children will have microcytic hypochromic anemia: their Hb < 11.5 g/L (Hb from 11.0-11.4 is mild anemia and in moderate anemia Hb is from 8.0-10.9 (WHO, 2011). The serum iron is below 60 mcg/dL (Elngar et al., 2021). The Ferritin level

   <12 µg/L for children in absence of infection (WHO, 2017). ( Appendix I).
3. They will be right handed.
4. They had no history of previous hand injuries, surgeries or other functional hand limitation.
5. All children will able to follow instructions and understand commands given during test procedures.
6. Their body mass index (BMI) will be ranged from 15.2 to 15.5 kg/m2 (WHO, 2007). (Appendix II).

Exclusion Criteria:

* Children will exclude if they have:

  1. Congenital or acquired deformity in the joints of upper limb.
  2. Unhealed fracture in upper limb bones.
  3. Systematic disease that cause anemia such as renal or hepatic failure or a history of bone disease.
  4. Blood transfusion within 3 months before measuring the hematological indices.
  5. Documented trauma in the previous 12 months in the muscle fibers, or those taking medication that affecting strength.
  6. Children begin with musculoskeletal problems or neurological disorders that affected their upper extremities
  7. Children who practice in any regular sport activities involving the upper extremities.8)

Ages: 5 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: eighty seven children from both sexes ranging in age from 5-6 years (thirty sex non-anemic children and fifty children with IDA (subdivided in to two equal groups. Group (I) 25 children with mild IDA and group (II) 25 children with moderate IDA). 2. They will be selected from the Outpatient Clinic of Pediatrics, Zagazig University Hospitals.
  3. The fifty anemic children will have microcytic hypochromic anemia:. for children aged 5-11 years old, Hb < 11.5 g/L (Hb from 11.0-11.4 is mild anemia and in moderate anemia Hb is from 8.0-10.9 (WHO, 2011). The serum iron is below 60 mcg/dL (Elngar et al., 2021). The Ferritin level <12 µg/L for children in absence of infection (WHO, 2017).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
measure tip to tip and tripod pinch strength | one year
  Baseline mechanical Pinch gauge (0-60 lb.) used to measure tip to tip and tripod pinch strength for all participated children
manual dexterity | one year
  Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2)
hemoglobin and serum iron levels | one year
  Fully automated blood cell counter (sysmex-Xs 800i) and AU 480-Chemistry auto-analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- the Outpatient Clinic of Pediatrics, Zagazig University Hospitals., Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No